CLINICAL TRIAL: NCT06408571
Title: Study on the Pathogenesis of Retinal Vascular Diseases Based on Body Fluid Metabolomics
Status: Enrolling by invitation | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20240202
Record Dates: First submitted 2024-03-21; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-02

CONDITIONS: Metabolomics; Retinopathy; Etiology
MeSH Terms: conditions — Retinal Diseases | interventions — Causality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients with retinal vein obstruction and diabetic retinopathy
  Interventions: Other: etiology
- Control group: Cataract surgery and vitrectomy patients

INTERVENTIONS:
Other: etiology — As an important part of systems biology, metabolomics mainly detects various metabolites in the sample. Different from nucleic acids, proteins and other biological macromolecules, the relative molecular weight of these metabolites is small, generally within 1000Da, such as amino acids, carboxylic acids, carbohydrates, alcohols, amines, lipids and other special substances. Through qualitative and quantitative analysis of all endogenous low molecular weight metabolites before and after pathophysiology or gene modification stimulation, metabolomics reveals the essential characteristics of life activities and metabolism of the body, and provides guidance for exploring the pathogenesis, early diagnosis, treatment and prognosis of diseases.
  Groups: Experimental group

SUMMARY:
Through the analysis of metabolites in body fluids (intraocular fluid, plasma) of patients with retinal vascular diseases (retinal vein occlusion, diabetic retinopathy), the possible pathogenesis of retinal vein occlusion was explored.

DETAILED DESCRIPTION:
1. Clinical data of patients with RVO and DR Were retrospectively studied to analyze their pathogenesis. 2. Metabolomic studies were conducted on body fluids (intraocular fluid and peripheral blood) of patients with RVO and DR And control group to find out the differences and find new targets for the prevention and treatment of RVO and DR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Confirmed diagnosis of retinal vein obstruction and diabetic retinopathy through ophthalmic specialist examination

Exclusion Criteria:

* Severe systemic diseases
* Pregnant and lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with RVO and DR Who were admitted to Zhongnan Hospital of Wuhan University from January 2018 to August 2023 (about 3600 cases)
Sampling Method: Non-Probability Sample
Enrollment: 3900 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Screening of prognostic markers and model validation | 1/12/2024-30/12/2024
  1. Surface markers and key molecules related to the study of diseases were screened out, and a biomarker model for assessing disease prognosis was established.
  2. Candidate differential molecules were screened through a training cohort, a Cox regression model was constructed, and the prognostic value of the model was verified in the test cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China